CLINICAL TRIAL: NCT04404504
Title: Smartphone-App Based Prediction of Large Vessel Occlusion in Suspected Stroke by Emergency Medical Service Using FAST-ED
Brief Title: Smartphone-App Based Prediction of Large Vessel Occlusion
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Martin Köhrmann, Prof. Dr. med., University Hospital, Essen
Other Study IDs: 18-8162
Record Dates: First submitted 2020-05-18; First posted 2020-05-27 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Acute Stroke
Keywords: Prehospital Triage
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this non-interventional study is to evaluate a German version of the triage stroke-score FAST-ED performed by ambulance service personnel in a pre-hospital setting using a smartphone app (Join-Triage, Allm).

DETAILED DESCRIPTION:
The emergency service of the city of Essen (NRW, Germany), which is organised by the Essen fire-department, will perform a prehospital triage stroke-score using a smartphone-app (Join-Triage, Allm) when referring patients with suspected stroke to the university clinic Essen. The triage stroke-score FAST-ED (Field Assessment Stroke Triage for Emergency Destination), as well as the expected time of arrival will be transmitted by an additional smartphone-app in advance of the arrival (Join, Allm). Patients will receive emergency workup to identify stroke etiology and presence of large vessel occlusion. Final diagnosis, presence of large vessel occlusion and type of revascularisation treatment will be registered. Sensitivity, specificity and further criteria for test quality will be calculated for the stroke triage by emergency service in field using the FAST-ED.

ELIGIBILITY:
All patients above the age of 18 with suspected acute stroke transferred to the university hospital Essen.

Inclusion criteria: suspected acute stroke, age above 18 years and a digitally transmitted FAST-ED by EMS prior to admission.

Exclusion criteria: Known symptom onset beyond 24 Hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with suspected acute stroke that are transferred by the Essen emergency service to the university hospital Essen shall be recruited
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Presence of large vessel occlusion | Baseline
  Acute stroke due to large vessel occlusion as measured by computed tomography angiography (CT-A)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Köhrmann, Prof. Dr., Study Director — University Hospital, Essen
Locations (1):
- University Hospital, Essen, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Frank B, Lembeck T, Toppe N, Brune B, Bozkurt B, Deuschl C, Nogueira RG, Dudda M, Risse J, Kill C, Forsting M, Kleinschnitz C, Kohrmann M. FAST-ED scale smartphone app-based prediction of large vessel occlusion in suspected stroke by emergency medical service. Ther Adv Neurol Disord. 2021 Nov 14;14:17562864211054962. doi: 10.1177/17562864211054962. eCollection 2021. PMID 34804205